CLINICAL TRIAL: NCT05498948
Title: Probiotic Mixture Supplementation (PMS) Promotes the Recovery of Patients After Heart Valve Replacement by Preventing Acute Gastrointestinal Injury (AGI)
Brief Title: PMS Promotes the Recovery of Patients After Heart Valve Replacement
Acronym: PMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Responsible Party: Principal Investigator, Wenbo Meng, Professor of Surgery, Hepatopancreatobiliary Surgery Institute of Gansu Province
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PMS
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Heart Valve Diseases
Keywords: Heart valve diseases; Probiotics; microbiomes; cardiac surgery
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic mixture (Experimental): Dietary Supplements: Probiotic mixture supplementation The Probiotic mixture supplementation contains Lactobacillus rhamnosus CMCC(B) P0028 ；Lactobacillus rhamnosus CMCC(B) P0029；Enterococcus faecium CMCC(B) P0030
  Interventions: Dietary Supplement: Probiotic mixture
- Placebo (Placebo Comparator): Dietary Supplement: Placebo The placebo product will be orally take.
  Interventions: Dietary Supplement: Probiotic mixture

INTERVENTIONS:
Dietary Supplement: Probiotic mixture — orally take .

SUMMARY:
Acute gastrointestinal injury (AGI) is related to poor outcomes in patients after heart valve replacement. The purpose of this study is to evaluate the effect of the probiotic mixture supplementation (PMS) in patients after heart valve replacement by preventing acute gastrointestinal injury (AGI).

DETAILED DESCRIPTION:
Patients with heart valve diseases often have chronic cardiac insufficiency. Accumulating evidence supports a relationship between the complexity and diversity of the gut microbiota and heart failure. Bacterial colonization and translocation of their toxins to the bloodstream due to altered intestinal permeability are directly correlated with systemic inflammation. The activation of pro-inflammatory pathways and chronic inflammation was hypothesized as a major contributing factor in the pathogenicity and progression of heart failure (HF) Patients undergoing heart valve replacement with cardiopulmonary bypass (CPB) are always complicated with gastrointestinal tract ischemia-reperfusion injury, which usually leads to AGI. AGI is related to poor outcomes of critically ill patients through many underlying mechanisms. It can leads to infectious complications, multiple organ dysfunction syndromes (MODS), and even death. On the other hand, the supply of probiotics, the good bacteria, is beneficial, despite still having a few controversial results. Therefore, it is important to carefully assess the efficacy of probiotics in the prevention of AGI and other complications in patients undergoing heart valve replacement surgery with CPB, as well as to evaluate the safety of its use.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe congestive heart failure (CHF) (NYHA functional class III to IV)
* Patients with heart valve diseases undergoing CPB cardiac surgery
* Age > 18 years and ≤ 70 years

Exclusion Criteria:

* Patients with severe low left ventricular function: LVEF ≤ 30%
* Patients with infective endocarditis
* Have received major gastrointestinal surgery (including gallbladder and appendectomy) within 5 years
* Inflammatory bowel disease (IBD), including ulcerative colitis, Crohn's disease, or colitis
* Acute gastroenteritis
* Clostridium difficile or Helicobacter pylori infection
* Chronic constipation
* Peptic ulcer
* Polyps in the stomach or intestines
* Gastrointestinal neoplasms
* Abdominal hernia
* Irritable bowel syndrome
* Acute or chronic cholecystitis, hepatitis
* Used antibiotics and probiotics in the past 1 month
* Patients used antidiarrheals, laxatives, or prebiotics within 1 week
* Pregnant or pregnant during follow-up
* Failure to give informed consent (e.g. severe cognitive impairment)
* The patient has been enrolled in other ongoing clinical trials

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-08-20 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
The AGI score | 1 month
  The AGI score of the patient within the 7th postoperative day was performed according to the European Society of critical care (2012) guidelines for AGI.
Intra-abdominal pressure (IAP) | 1 month
  We defined it as the maximum value of intra-abdominal pressure within 7 days after surgery
Characteristics of gut microbiomes | 1 month
  Feces are collected with sterilized 2 ml tubes and frozen at -80 °C until DNA extraction, preparing for microbe analysis

SECONDARY OUTCOMES:
Return time of bowel sounds | 1 month
  The return time of bowel sounds will be evaluated morning and evening
Number of bowel sounds | 1 month
  The number of bowel sounds will be evaluated morning and evening
First defecation time | 1 month
  The time to the first defecation will be asked morning and evening after surgery
Bristol Stool Form Scale score | 1 month
  Bristol Stool Form Scale is a medical aid designed to classify the form of stool with 7 levels
Proportion of cocci and bacilli in feces | 1 month
  The first feces will be collected in sterile containers for the tertial smear
Procalcitonin (PCT) | 1 month
  Blood samples will be collected on the 1st and 3rd days after operation, for analyses of the PCT
Interleukin-6 | 1 month
  Blood samples will be collected on the 1st and 3rd days after operation, for analyses of the Interleukin-6
Interleukin-10 | 1 month
  Blood samples will be collected on the 1st and 3rd days after operation, for analyses of the Interleukin-10
High sensitivity troponin(hs TnI) | 1 month
  Blood samples will be collected on the 1st and 3rd days after operation, for analyses of the hs TnI
N-terminal precursor brain natriuretic peptide(NT-ProBNP) | 1 month
  Blood samples will be collected on the 1st and 3rd days after operation, for analyses of the NT-ProBNP
Trimethylamine oxide(TMAO) | 1 month
  Blood samples will be collected on the 1st and 3rd days after operation, for analyses of the TMAO
Intestinal fatty acid-binding protein (IFABP) | 1 month
  Blood samples will be collected on the 1st and 3rd days after operation, for analyses of the IFABP
Left ventricular ejection fraction (LVEF) | 1 month
  Measure the LVEF on the 1st and 3rd days after operation by echocardiographic examinations

CONTACTS AND LOCATIONS:
Overall Officials: Wenbo Meng, M.D. Ph.D,, Principal Investigator — LanZhou University
Locations (1):
- Hepatopancreatobiliary Surgery Institute of Gansu Province, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No
If patients permitted

REFERENCES:
- [Result] Pasini E, Aquilani R, Testa C, Baiardi P, Angioletti S, Boschi F, Verri M, Dioguardi F. Pathogenic Gut Flora in Patients With Chronic Heart Failure. JACC Heart Fail. 2016 Mar;4(3):220-7. doi: 10.1016/j.jchf.2015.10.009. Epub 2015 Dec 9. PMID 26682791
- [Result] Chen Y, Zhang F, Ye X, Hu JJ, Yang X, Yao L, Zhao BC, Deng F, Liu KX. Association Between Gut Dysbiosis and Sepsis-Induced Myocardial Dysfunction in Patients With Sepsis or Septic Shock. Front Cell Infect Microbiol. 2022 Mar 14;12:857035. doi: 10.3389/fcimb.2022.857035. eCollection 2022. PMID 35372123
- [Derived] Yang X, Liu R, An Z, Li B, Lin Y, Li Y, Song B, Yuan J, Meng W, Waydhas C. Probiotic mitigates gut hypoperfusion-associated acute gastrointestinal injury in patients undergoing cardiopulmonary bypass: a randomized controlled trial. BMC Med. 2025 Apr 23;23(1):238. doi: 10.1186/s12916-025-04082-2. PMID 40264088